CLINICAL TRIAL: NCT06167005
Title: National Introduction of One Anastomosis Gastric Bypass in the UK National Bariatric Surgery Registry
Status: Completed | Type: Observational
Sponsor: British Obesity and Metabolic Surgery Society (Other Government)
Responsible Party: Principal Investigator, Andrew Currie, Andrew Currie, British Obesity and Metabolic Surgery Society
Other Study IDs: 0001
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- One anastomosis gastric bypass
  Interventions: Procedure: Primary bariatric-metabolic surgery
- Roux en y gastric bypass
  Interventions: Procedure: Primary bariatric-metabolic surgery
- Sleeve gastrectomy
  Interventions: Procedure: Primary bariatric-metabolic surgery
- Adjustable gastric band
  Interventions: Procedure: Primary bariatric-metabolic surgery

INTERVENTIONS:
Procedure: Primary bariatric-metabolic surgery — Primary bariatric-metabolic surgery

SUMMARY:
This study is investigating a newer surgical procedure called one-anastomosis gastric bypass (OAGB) used for treating obesity within the National Health Service (NHS). We want to understand how well this surgery works and its effects on patients' health. We'll look at data from adults who had this surgery, tracking everything from before the operation to after they go home and comparing to other types of operation for weight loss. We'll check for any problems during or after surgery, how long they stay in the hospital, and how much weight they lose. We're also interested in seeing if other health issues related to obesity get better. By doing this, we hope to learn more about how effective and safe this surgery is and how it's being used in hospitals across the country

DETAILED DESCRIPTION:
Recent reporting from the International Federation for Surgery for Obesity (IFSO) Registry report that the three most common metabolic surgery procedures are sleeve gastrectomy (SG), Roux-en-y gastric bypass (RYGB) and one-anastomosis gastric bypass (OAGB)[1]. Introduced by Rutledge in 1997[2], OAGB is now increasing being used in bariatric practice. Recent network meta-analysis indicates OAGB may offer comparable weight loss whilst minimising complications[3]. Literature published from both the IFSO Registry and the Israeli National Registry indicate increased use of OAGB in the surgical treatment of obesity[1, 4].

The safe introduction of new surgical procedures can be confounded by learning effects for both operative technique and perioperative care practices[5]. No study has yet considered the introduction of OAGB at a population or national registry level.

The aim of the study is to study the introduction of OAGB into NHS practice in the national bariatric surgery registry.

Study population: Adult patients undergoing surgery for obesity using one-anastomosis gastric bypass Exclusions: Paediatric cases

Data All patient undergoing OAGB operations within the NBSR - pre-operative, intra-operative and postoperative data as described below

Outcome measures Perioperative outcomes Complications Return to theatre Length of stay Percentage of OAGB practice as a proportion of total bariatric surgery practice at individual hospitals

Longer term outcomes Total body weight loss Excess weight loss Remission of comorbidities

References

1. Welbourn R, Hollyman M, Kinsman R, Dixon J, Cohen R, Morton J, et al. Bariatric-Metabolic Surgery Utilisation in Patients With and Without Diabetes: Data from the IFSO Global Registry 2015-2018. Obes Surg. 2021 Feb 27. PubMed PMID: 33638756. Epub 2021/02/28.
2. Rutledge R. The mini-gastric bypass: experience with the first 1,274 cases. Obes Surg. 2001 Jun;11(3):276-80. PubMed PMID: 11433900. Epub 2001/07/04.
3. Currie AC, Askari A, Fangueiro A, Mahawar K. Network meta-analysis of metabolic surgery procedures for the treatment of obesity and diabetes. Obes Surg. In Press.
4. Kaplan U, Romano-Zelekha O, Goitein D, Keren D, Gralnek IM, Boker LK, et al. Trends in Bariatric Surgery: a 5-Year Analysis of the Israel National Bariatric Surgery Registry. Obes Surg. 2020 May;30(5):1761-7. PubMed PMID: 32008257. Epub 2020/02/03.
5. Dimick JB, Sedrakyan A, McCulloch P. The IDEAL Framework for Evaluating Surgical Innovation: How It Can Be Used to Improve the Quality of Evidence. JAMA Surg. 2019 Jun 5. PubMed PMID: 31166583. Epub 2019/06/06.

ELIGIBILITY:
Inclusion Criteria:

* All primary bariatric metabolic surgeries performed between January 2009 and December 2019

Exclusion Criteria:

* Individuals under 18 years of age, those undergoing revisional surgery (defined as conversion to another bariatric procedure), or gastric balloon insertion as the sole treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing primary bariatric metabolic surgery within the UK National Bariatric Surgery Registry
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity | 30 day
Weight loss | 12 month

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Welbourn R, Hollyman M, Kinsman R, Dixon J, Cohen R, Morton J, Ghaferi A, Higa K, Ottosson J, Pattou F, Al-Sabah S, Anvari M, Himpens J, Liem R, Vage V, Walton P, Brown W, Kow L. Bariatric-Metabolic Surgery Utilisation in Patients With and Without Diabetes: Data from the IFSO Global Registry 2015-2018. Obes Surg. 2021 Jun;31(6):2391-2400. doi: 10.1007/s11695-021-05280-6. Epub 2021 Feb 27. PMID 33638756
- [Background] Rutledge R. The mini-gastric bypass: experience with the first 1,274 cases. Obes Surg. 2001 Jun;11(3):276-80. doi: 10.1381/096089201321336584. PMID 11433900
- [Background] Currie AC, Askari A, Fangueiro A, Mahawar K. Network Meta-Analysis of Metabolic Surgery Procedures for the Treatment of Obesity and Diabetes. Obes Surg. 2021 Oct;31(10):4528-4541. doi: 10.1007/s11695-021-05643-z. Epub 2021 Aug 7. PMID 34363144
- [Background] Kaplan U, Romano-Zelekha O, Goitein D, Keren D, Gralnek IM, Boker LK, Sakran N. Trends in Bariatric Surgery: a 5-Year Analysis of the Israel National Bariatric Surgery Registry. Obes Surg. 2020 May;30(5):1761-1767. doi: 10.1007/s11695-020-04426-2. PMID 32008257
- [Background] Dimick JB, Sedrakyan A, McCulloch P. The IDEAL Framework for Evaluating Surgical Innovation: How It Can Be Used to Improve the Quality of Evidence. JAMA Surg. 2019 Aug 1;154(8):685-686. doi: 10.1001/jamasurg.2019.0903. No abstract available. PMID 31166583
- [Derived] Currie AC, Askari A, Parmar C, Byrne J, Ahmed AR, Pring CM, Khan OA, Small PK, Mahawar K. National introduction of one-anastomosis gastric bypass in the UK National Bariatric Surgery Registry: a cohort study. Int J Surg. 2024 Dec 1;110(12):7404-7413. doi: 10.1097/JS9.0000000000002005. PMID 39311895